CLINICAL TRIAL: NCT05835128
Title: A Multicentric Prospective Study: Assessment of Pulmonary Long-term Sequelae of Coronavirus Disease 2019 (COVID-19) Pneumonia With Chest Computed Tomography and Pulmonary Function Tests
Brief Title: Assessment of Long-term Sequelae of Coronavirus Disease 2019 (COVID-19) Pneumonia With Chest CT and Pulmonary Function Tests
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centro Hospitalar Universitario do Algarve (Other)
Collaborators: Universidade do Algarve (Other)
Responsible Party: Principal Investigator, Mónica Diniz, MD, Principal Investigator, Centro Hospitalar Universitario do Algarve
Other Study IDs: UAIF 96/2020
Record Dates: First submitted 2023-04-25; First posted 2023-04-28 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: COVID-19 Pneumonia; Sequelae of; Infection; Respiratory Function Impaired; SARS CoV 2 Infection; SARS-CoV 2 Pneumonia
Keywords: COVID-19; Tomography; Infections, Viral; Respiratory Tract Infections; Virus Disease; Coronavirus Infections; Infections; Lung Diseases; RNA virus infections; Respiratory tract diseases; Chest CT; Reduced dose chest CT; Lung CT; coronaviridae infections; lung sequela; pneumonia; respiratory function tests; follow-up studies; multicentric studies; prospective studies
MeSH Terms: conditions — Infections; Respiratory Insufficiency; COVID-19; Virus Diseases; Respiratory Tract Infections; Coronavirus Infections; Lung Diseases; RNA Virus Infections; Respiratory Tract Diseases; Coronaviridae Infections; Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective multicentric study is to evaluate the presence of long-term pulmonary sequelae in patients who had required hospitalization for treating COVID-19 pneumonia, trough chest CT and pulmonary function tests (PFT).

Secondly we would like to evaluate the possible correlation between the chest CT findings and pulmonary function tests pre-existing co-morbidities and type of therapy used during hospitalization.

DETAILED DESCRIPTION:
The investigators will invite to participate in this study patients who had been hospitalized with positive test for severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) , namely with positive reverse transcription polymerase chain reaction or positive rapid antigen test, and with respiratory insufficiency (at admission or developed during hospital stay), or with viral pneumonia documented with thorax x-ray or Chest CT, during the period between march 2020 and march 2022.

Patients who agree to participate and sign the informed consent will be enrolled in the study.

Participants will be evaluate in two different periods: approximately 4 to 6 months after hospital discharge and approximately 12 to 14 months after hospital discharge.

The first evaluation includes a physical examination at medical post-COVID-19 consultation, pulmonary function tests and reduced dose chest CT.

The second evaluation includes a physical examination at medical post-COVID-19 consultation, and will include reduced dose chest CT and pulmonary function tests only if there were significative findings on those exams on the first evaluation, or if there are any clinical significative findings at the present moment.

All the evaluations must respect the following time intervals: the pulmonary function tests and the chest CT will be done within a 6 week maximum interval of each other, and both of these examinations will be done within a 8 week maximum interval regarding the clinical evaluation.

Demographic and clinical data will be collected by qualified clinical study staff (i.e., by physicians who conduct the post-COVID-19 medical consultation) and the patient will given the EuroQol 5 Dimension 5 Level questionnaire (EQ-5D-3L) to assess the health status.

The reduced dose Chest CT will be obtained with the patient in a supine position and with breath-holding following inspiration, in a spiral acquisition mode with a 1 ,5 mm slice thickness and the images will be reviewed by four senior radiologist blinded to clinical and respiratory functional tests results.

The pulmonary function tests will be interpreted according to the American Thoracic Society and European Respiratory Society guidelines 2022. The parameters measured included the forced expiratory flow between 25% and 75% of forced vital capacity (FVC), forced expiratory volume (FEV1), FVC/FEV1, vital capacity, total lung capacity, residual volume and the diffusing capacity of lung for carbone monoxide (DLCO), DLCO/Alveolar Volume (AV).

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years old of age;
* positive SARS-CoV-2 reverse transcription-polymerase chain reaction on a nasopharyngeal and/or oropharyngeal swab or positive SARS-CoV-2 rapid antigen test
* hospitalization in one of two hospitals of our institution (university center) in consequence of SARS-CoV-2 related disease between march of 2020 and march of 2022 and having :
* respiratory insufficiency when admitted or developing after admission or image documented viral pneumonia ;
* at least one thorax x-ray or lung CT acquired during the hospitalization period

Exclusion Criteria:

* previous lung cancer
* previous intersticial lung disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted in two Portuguese hospitals from the same institution (university center). Patients will be recruited from the follow -up Post-COVID-19 medical consultations. All patients attending these follow- up consultations will be invited to participate and enrolled if they agree to sign the written informed consent (following the ethics committee protocol).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of structural lung sequelae after COVID-19 pneumonia | 12 -14 months
  evaluate the presence of lung structural sequelae with chest CT
Prevalence of functional lung impairment after COVID-19 pneumonia | 12 -14 months
  evaluate the presence of impaired PFT after COVID-19 pneumonia
Association between chest CT findings and PFT impairment after COVID-19 pneumonia | 12-14 months
  evaluate the possible correlation between the presence of pulmonary structural alterations on chest CT and the presence of impaired PFT

SECONDARY OUTCOMES:
Prevalence of structural lung sequelae after COVID-19 pneumonia | 4-6 months
  evaluate the presence of lung structural sequelae with chest CT
Prevalence of functional lung impairment after COVID-19 pneumonia | 4-6 months
  evaluate the presence of impaired PFT after COVID-19 pneumonia
Association between chest CT findings and PFT impairment after COVID-19 pneumonia | 4-6 months
  evaluate the possible correlation between the presence of pulmonary structural alterations on chest CT and the presence of impaired PFT
Association between chest CT findings after COVID-19 pneumonia and therapy used during hospitalization | 4-6 months
  to evaluate if there is any association between the presence of lung structural sequelae on chest CT and the different treatments used during hospitalization (corticotherapy, oxygen therapy, mechanical ventilation)
Association between chest CT findings after COVID-19 pneumonia and therapy used during hospitalization | 12-14 months
  to evaluate if there is any association between the presence of lung structural sequelae on chest CT and the different treatments used during hospitalization (corticotherapy, oxygen therapy, mechanical ventilation)
Association between chest CT findings after COVID-19 pneumonia and pre-existing co-morbidities | 4-6 months
  to evaluate if there is any association between the presence of lung structural sequelae on chest CT and pre-existing co-morbidities (diabetes, asthma, hypertension, dyslipidaemia, obesity, chronic obstructive pulmonary disease, cigarette smoking, heart disease and kidney disease)
Association between chest CT findings after COVID-19 pneumonia and pre-existing co-morbidities | 12 -14 months
  to evaluate if there is any association between the presence of lung structural sequelae on chest CT and pre-existing co-morbidities (diabetes, asthma, hypertension, dyslipidaemia, obesity,, chronic obstructive pulmonary disease, cigarette smoking, heart disease and kidney disease)

CONTACTS AND LOCATIONS:
Overall Officials: Mónica Diniz, MD, Principal Investigator — unafilliated; Castro Miguel, MD, Principal Investigator — Centro Hospitalar Universitário do Algarve/Polo de Portimão
Locations (2):
- Portugal (2):
  - Hospital de Faro (CHUA), Faro
  - Hospital de Portimâo (CHUA), Portimão

IPD SHARING:
Plan to Share IPD: Undecided